CLINICAL TRIAL: NCT01676350
Title: Intraosseous Access in the Emergency Department for Patients With Failed Attempts at Intravenous Access: A Randomized Trial Examining Resource Utilization and Patient Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: WellSpan Health (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 299341
Record Dates: First submitted 2012-08-28; First posted 2012-08-30 (Estimated); Results first posted 2022-03-08 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Difficult Peripheral IV Access
Keywords: Intraosseous (IO) vascular access

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of care (No Intervention): If you are assigned to this group, ultrasound-guided IV will be used to obtain vascular access.
- IO access using EZ-IO® (Experimental): If you are assigned to this group, you will receive an IO line in the humeral head of the shoulder. IO lines are placed using an FDA-approved device called an EZ-IO®.
  Interventions: Procedure: IO access using EZ-IO®

INTERVENTIONS:
Procedure: IO access using EZ-IO® — IO line placed using an FDA-approved device called an EZ-IO®.
  Other Names: EZ-IO®
  Arms: IO access using EZ-IO®

SUMMARY:
By doing this study, the investigators hope to learn whether patients with difficult to obtain IV access who are treated with IO access are more satisfied with their care and have better outcomes. The investigators are specifically studying the time difference between groups and the difference in the number of attempts required to obtain vascular access and begin to treat with fluids and medications. The study will also measure patient satisfaction and procedural pain, the frequency of central line placement, the length of stay in the hospital and emergency department, and adverse events to intravascular access to determine whether IO access can improve these measures.

The investigators hypothesize that the use of a protocol utilizing an IO device for select patients with failed IV access will reduce the time requirements to obtain vascular access, reduce the number of attempts needed to obtain IV access, reduce the ED LOS, and have no negative impact on patient satisfaction compared to the current ED practices.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Hemodynamically stable
3. Speaks English
4. Able to consent
5. Has difficult IV access

Exclusion Criteria:

1. Patients who are younger than 18 years of age, b) lack English fluency c) are unable to give informed consent d) require immediate central venous access e) have a history of osteomyelitis in the only target location of IO access f) have a fracture in the bone of the only target IO site g) have received an IO in the last 24 hours of the only target site h) are allergic to lidocaine i) pregnant or j) require a contrast CT scan as part of their ED care will be excluded.

While pregnant patients may benefit from rescue access the use of lidocaine to anesthetize the medullary space has not been studied in this population.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erik Kochert, MD, Principal Investigator — York Hospital
Locations (2):
- United States (2):
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - York Hospital, York, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Groups:
- &Apos;IO Access Using EZ-IO®: If you are assigned to this group, you will receive an IO line in the humeral head of the shoulder. IO lines are placed using an FDA-approved device called an EZ-IO®.
  IO access using EZ-IO®: IO line placed using an FDA-approved device called an EZ-IO®.
Period: Overall Study
Arm/Group | Standard of Care | &Apos;IO Access Using EZ-IO®
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Standard of Care: Standard of care
- IO Access: IO access
- Total: Total of all reporting groups
Arm/Group | Standard of Care | IO Access | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 10 | 19
  >=65 years | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 8 | 15
  Male | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Time to Successful Placement of a Functioning USGIV/IO
Time Frame: at time of vascular access
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Standard of Care | &Apos;IO Access Using EZ-IO®
Number analyzed (Participants) | 11 | 8
seconds | 163.7 (177.9) | 67.3 (98.5)

2. Primary Outcome: Number of Successful Placements
Time Frame: at time of vascular access
Measure: Number; unit: successful placements
Arm/Group | Standard of Care | IO Access Using EZ-IO®
Number analyzed (Participants) | 11 | 11
successful placements | 11 | 8

ADVERSE EVENTS:
Arm/Group | Standard of Care | &Apos;IO Access Using EZ-IO®
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No